CLINICAL TRIAL: NCT06905769
Title: Effects of Aquatic Therapy Versus Neuro-dynamic Technique for the Treatment of Carpal Tunnel Syndrome Patient: A Randomized Clinical Trial
Brief Title: Effects of Aquatic Therapy Versus Neuro-dynamic Technique for the Treatment of Carpal Tunnel Syndrome Patient
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/787
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Aquatic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Therapy (Experimental)
  Interventions: Combination Product: Aquatic Therapy
- Neuro-Dynamic Technique (Experimental)
  Interventions: Diagnostic Test: Neuro-Dynamic Technique

INTERVENTIONS:
Combination Product: Aquatic Therapy — Group A was treated with Aquatic Therapy for 30-45 minutes for 3 sessions per week for 8 weeks . Patient should Seated .Therapist will standing or seated beside the patient Therapist Perform gentle stretching on wrist, hand, and finger joints. Exercises to improve range of motion and reduce stiffness. Then perform aquatic therapy for 10 minutes. Therapist instruct patients hands in bath tube. Water temperature 88°F - 94°F (31°C - 34°C).Water depth is Waist-deep or deeper depending on patient comfort
  Arms: Aquatic Therapy
Diagnostic Test: Neuro-Dynamic Technique — Group B (Neuro-Dynamic Technique) Group B was treated with Neuro-Dynamic Technique for 15 minutes 3 sessions per week for 8 weeks. Patient should Seated or supine with the affected hand relaxed. Therapist will standing or seated beside the patient. Techniques Time duration is 3 minutes for each technique. wrist distraction 3 sets for 3 minute rhythmic and gentle stretching of the transverse carpel ligament Release of palmar fascia gliding of finger flexor tendons release of upper forearm muscle and fascia.
  Arms: Neuro-Dynamic Technique

SUMMARY:
Carpal Tunnel Syndrome (CTS) is a common neurological disorder due to entrapment of median nerve which runs from the forearm into the hand through a tunnel, compressed or pinched due to anatomical factors, such as a narrow carpal tunnel. Widespread condition that affects 3-6% of the general population worldwide. Carpal Tunnel Syndrome (CTS) a prevalent and debilitating condition leading to disability despite optimal interventions to rehabilitation that aimed to reducing pain and improving neural function status in Carpal Tunnel Syndrome Patients .

DETAILED DESCRIPTION:
This study investigates the additional benefits of Aquatic Therapy and Neuro-dynamic Technique in Carpal Tunnel Syndrome Patients .The researcher employs a randomized controlled trial methodology. Participants are divided into two groups: one receiving Aquatic Therapy, and the other receiving Neuro-dynamic Technique.

Outcomes are assessed over an 8-week period, focusing on pain levels and neural function restoration and grip strength. The significance of this study lies in its potential to enhance current treatment protocols, offering a more effective, intervention to alleviate symptoms and improve the quality of life, neural restoration for those suffering Carpal Tunnel Syndrome (CTS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild-to-moderate carpal tunnel syndrome by Neuromuscular Physician
* Participants who presented with unilateral CTS with symptoms reported up to 3 months
* Male and female
* Aged 18 years or older

Exclusion Criteria:

* Patients with non-specified stage of CTS,median nerve entrapment in TOS, Cervical Radiculpathy
* Participants presents with co-morbidities,Hx of CTS (e.g., pregnancy, diabetes, trauma, congenital disorders, obesity, post-surgical release, and hypothyroidism)
* Cardiovascular disease, thenar muscle atropy"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE (NPRS) | 12 Months
  The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine" or "worst pain imaginable". The NPRS is a valid and reliable scale to measure pain intensity. NPRS demonstrates strong correlation validity with other established pain measurement scales, making it a reliable tool for clinical assessments.
Boston Carpal Tunnel Questionnaire (BCTQ) | 12 Months
  The questionnaire has been designed to evaluate Assess the severity of CTS symptoms and functional impairment. The total number of questions is 19, total score is 95(sum of 2 subscales) in the BCTQ. Symptom Severity Scale (SSS): 11 items assessing the severity of CTS symptoms, such as numbness, tingling, and pain. Functional Status Scale (FSS) 8 items evaluating the impact of CTS on daily activities, such as grasping, gripping, an carrying. Symptom Severity Scale (SSS): Scores range from 1-5, with higher scores indicating more severe symptoms Functional Status Scale (FSS): Scores range from 1-5, with higher scores indicating greater functional impairment .Reliability 0.95% and Validity 0.80%.
  Interpretation
  Symptom Severity Scale (SSS) Mild symptoms: 1-2 Moderate symptoms: 2-3 Severe symptoms: 3-4 Very severe symptoms: 4-5
Grip Strength | 12 Months
  Digital Hand Dynamometer is a device used to measure grip strength, which is the force exerted by the hand when grasping an object. Hand Dynamometer units of measurement typically represents the maximum grip strength measured in units Kilograms (kg),Pounds (lb) And Newtons (N). Standard-range dynamometers: 0-100 kg (0-220 lb).
  Normal Values for Grip Strength Adult Men: 35-55 kg Adult Women: 20-35 kg
  Interpretation
  Mild Weakness: 10-20% below normal range. Moderate Weakness: 20-40% below normal range. Severe Weakness: 40-60% below normal range. Profound Weakness: More than 60% below normal range."

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University CRC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No